CLINICAL TRIAL: NCT03513432
Title: Influence of Beer on Gut Microbiota and Biochemical Outcomes: Alcohol Impact.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MICROAL
Record Dates: First submitted 2018-04-12; First posted 2018-05-01 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Gut microbiota; Beer; Alcohol; Cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Beer; Ethanol

STUDY DESIGN:
Intervention Model Description: This is a three-arm parallel-group, randomized controlled study to evaluate the effect of consumption of beer with or without alcohol (5.20 %, 0.45 % and 0.00 %), during 4 weeks, on healthy individuals.
  The study will focus on the effects of beer on microbiota and biochemical biomarkers in healthy human volunteers.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beer with 5.20 % alcohol (Experimental): 330 ml beer (5.20 % alcohol)/day
  Interventions: Dietary Supplement: Beer with 5.20 % alcohol
- Non-alcoholic beer with 0.45 % alcohol (Experimental): 330 ml non-alcoholic beer (0.45 % alcohol)/day
  Interventions: Dietary Supplement: Non-alcoholic beer with 0.45 % alcohol
- Non-alcoholic beer with 0.00 % alcohol (Experimental): 330 ml non-alcoholic beer (0.00 % alcohol)/day
  Interventions: Dietary Supplement: Non-alcoholic beer with 0.00 % alcohol

INTERVENTIONS:
Dietary Supplement: Beer with 5.20 % alcohol — 330 ml beer (5.20 % alcohol)/day during 4 weeks
  Arms: Beer with 5.20 % alcohol
Dietary Supplement: Non-alcoholic beer with 0.45 % alcohol — 330 ml non-alcoholic beer (0.45 % alcohol)/day during 4 weeks
  Arms: Non-alcoholic beer with 0.45 % alcohol
Dietary Supplement: Non-alcoholic beer with 0.00 % alcohol — 330 ml nonalcoholic beer (0.00 % alcohol)/day during 4 weeks
  Arms: Non-alcoholic beer with 0.00 % alcohol

SUMMARY:
Our aim is to assess the effects of moderate consumption of beer and non-alcoholic beer on gut microbiota and biochemical biomarkers in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adult men (18-65 years);
* Healthy volunteers free of chronic diseases with relevant effect on gastrointestinal system;
* Without a diagnosis of any digestive disease including functional bowel disorders such as IBS;
* Moderate alcohol consumers;
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Documented cardiovascular disease (ischaemic heart disease - angina or recent or old myocardial infarction or previous or cerebral vascular accident, peripheral vascular disease);
* With diabetes or other relevant metabolic diseases;
* With any known infectious diseases, namely infections with HIV, Hepatitis B or C virus;
* Intake of antibiotics in the last 4 weeks and laxatives in the last 2 weeks;
* Subjects with history of drug, alcohol or other substances abuse.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in intestinal microbiota from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)

SECONDARY OUTCOMES:
Changes in fasting serum total cholesterol from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
Changes in fasting serum triglycerides from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
Changes in fasting serum cHDL from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
Changes in fasting serum cLDL from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
Changes in Homeostasis Model Assessment-Insulin Resistance (HOMA-IR) from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
Changes in body mass index from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
  Weight and height will be combined to report BMI in kg/m^2.
Changes in total body fat mass from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)
Changes in fasting serum LPS levels from baseline | at visit 1 (after 1-week run-in period) and at visit 2 (after 4-week intake period)

CONTACTS AND LOCATIONS:
Overall Officials: Conceição Calhau, PhD, Principal Investigator — NOVA Medical School
Locations (1):
- Faculdade de Ciências Médicas da Universidade NOVA de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: Undecided